CLINICAL TRIAL: NCT07135219
Title: An Open-Label Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Preliminary Clinical Activity of Cizutamig in Patients With Immunoglobulin A Nephropathy
Brief Title: A Study of Cizutamig in Patients With Immunoglobulin A Nephropathy
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CND106-PUFH-1
Record Dates: First submitted 2025-08-01; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Immunoglobulin A Nephropathy (IgAN)
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A study of cizutamig in patients with immunoglobulin A nephropathy (Experimental): Experlmental: Cizutamig intravenous intervention
  Interventions: Drug: Biological: cizutamig

INTERVENTIONS:
Drug: Biological: cizutamig — Cizutamig will be dosed according to the protocol.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, PK, PD, immunogenicity, and preliminary clinical activity of cizutamig in patients with IgAN.

DETAILED DESCRIPTION:
An Open-Label Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Preliminary Clinical Activity of Cizutamig in Patients with Immunoglobulin A Nephropathy

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age at the time of signing the informed consent form (ICF).
* Biopsy-confirmed IgAN as specified in the protocol.
* 24-hour urine protein excretion ≥1.0 g/day or 24-hour urine protein to creatinine ratio (uPCR) ≥0.75 g/g .
* Inadequate response to ≥1 of the therapies defined in the protocol.
* eGFR >30 mL/min/1.73m2.

Exclusion Criteria:

* Inadequate clinical laboratory parameters at Screening.
* Receipt of or inability to discontinue any of the following excluded therapies as specified in the protocol.
* Receipt of live vaccine within 4 weeks prior to Screening.
* MEST-C score of T2 from the Oxford IgAN classification schema. If MEST-scoring was not performed, the presence of >50% tubular atrophy/interstitial fibrosis is exclusionary.
* Rapidly progressing glomerulonephritis with eGFR reduction ≥50% within 12 weeks of Screening.
* Secondary IgAN (eg, chronic liver disease, celiac disease, HIV).
* History of IgA vasculitis.
* Presence of any concomitant autoimmune disease .
* History of progressive multifocal leukoencephalopathy.
* History of primary immunodeficiency or a hereditary deficiency of the complement system.
* Central nervous system (CNS) disease .
* Presence of 1 or more significant concurrent medical conditions per investigator judgment.
* Diagnosis or history of malignant disease within 5 years prior to Screening.
* Tonsillectomy within 24 weeks prior to Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Baseline up to 52 weeks
  Incidence and severity of TEAEs through end of study：
  1. Incidence and severity of treatment-emergent adverse events through end of study
  2. Changes from baseline in vital signs, ECG, and laboratory assessments through end of study

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No